CLINICAL TRIAL: NCT03606759
Title: Evaluation of the Efficacy of the Individually Adjusted Therapy Scale (ATI) on the Addiction Severity of Patients in Treatment for a Substance Use Disorder or a Behavioral Addiction. A Multicenter Randomized Controlled Trial (AjusT)
Brief Title: Evaluation of the Efficacy of the Individually Adjusted Therapy Scale (ATI) on the Addiction Severity
Acronym: AjusT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2014/43
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Addictive Behavior; Substance-Related Disorders
Keywords: Addiction; High-risk relapse situation; Craving; Individual cues; Individually tailored treatment
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traitment as usual adjusted on ATI information (Experimental): Assessments with a multidisciplinary team (doctors, nurses, psychologists, psychiatrists, social workers) once a week during 3 months.
  Interventions: Procedure: Weekly assessment ajusted
- Traitment as usual (Active Comparator): Assessments with a multidisciplinary team (doctors, nurses, psychologists, psychiatrists, social workers) once a week during 3 months.
  Interventions: Procedure: Weekly assessment

INTERVENTIONS:
Procedure: Weekly assessment — Weekly assessment during 3 months :
  Severity of addiction (Addiction Severity Index, ASI) Mini International Neuropsychiatric Interview, MINI Craving intensity (BILAN-7 jours) Individual cues of each participant (QSA) Substance use and gambling (BILAN-7 jours)
  Arms: Traitment as usual
Procedure: Weekly assessment ajusted — Weekly assessment during 3 months :
  Severity of addiction (Addiction Severity Index, ASI) Mini International Neuropsychiatric Interview, MINI Craving intensity (BILAN-7 jours) Individual cues of each participant (QSA) Substance use and gambling (BILAN-7 jours) Individually Adjusted Therapy scale (ATI)
  Arms: Traitment as usual adjusted on ATI information

SUMMARY:
The management of the craving is a key element in addiction treatment as the craving is linked to the probability of relapse. Several cues could induce the craving, some generic substance-induced cues or addictive behavior-related cues (e.g. gambling-related cues), and also some more subject-specific cues. The awareness of the craving intensity and its individual cues for each patient will allow the clinician to tailor a better treatment. The aim of this study is to evaluate the efficacy of a program based on an Individually Adjusted Therapy scale added to a treatment as usual for the treatment of addiction.

DETAILED DESCRIPTION:
Addiction is one of the most prevalent psychiatric disorders in general population. In the DSM-5, substance abuse and substance dependence have been combined into a single substance use disorder and gambling disorder is now reclassified in the new substance-related and addictive disorders category. Moreover, a criterion assessing the craving has been added. The management of craving is an important focus of addiction treatment as craving is often linked to relapse. Several cues could precipitate the craving. Some of them are substance-related or gambling-related, some other are more person-specific. Recent studies have revealed that those "individual cues" are highly predictive of craving and relapse, and suggest that they are involved in addiction chronicity. The awareness of these cues and the intensity of the craving are important to tailor a better treatment adapted to the patient's need in order to prevent relapse. The aim of this study is to evaluate the efficacy of a program that includes an Individually Adjusted Therapy scale (ATI) to help the clinician to modulate the level of care regarding of the patient's risk of relapse (based on cues, intensity and frequency of the craving). The study will consist in a randomized controlled trial comparing 2 groups of participants that are seeking treatment for substance use disorder (alcohol, opiates, tobacco, cannabis, cocaine or any other substance) or behavioral addiction in an outpatient addiction clinics in France (four inclusion sites).

All the participants will be assessed with several questionnaires that evaluate the history and the severity of addiction.

ELIGIBILITY:
Inclusion criteria:

* 18 years old or older
* Meet DSM-5 substance use disorder diagnosis for at least one substance (alcohol, tobacco, cannabis, opiates, cocaine or any other substance) use disorder or behavioral addiction (gambling, screens, video games, food addiction, sex addiction, compulsive purchases), currently not stabilized
* Seek treatment for this a substance use disorder or behavioral addiction
* Beginning (or re-initiating) multi-month outpatient care for this disorder in one of the inclusion centres.
* Ability to identify a priority substance/behavior, as main object of treatment, in case of simultaneous treatment on several addictions
* Beneficiary of the French Social Security system
* Give an informed consent to participate

  o Exclusion criteria:
* Severe physical or psychiatric or addictologic condition that prevents an outpatient treatment
* Severe physical or psychiatric condition that prevents to complete the assessment
* Addictive disorder that requires several treatment for several substance use disorder simultaneously
* Difficulty to understand and to write French
* Could not be reachable by phone
* Participate to another study that prevents to participate to another research
* Prisoner
* Person under law protection
* Person under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Craving intensity (BILAN-7 jours) | 3 month
  Craving intensity measured by the difference in craving intensity score at baseline and 3-month follow-up

SECONDARY OUTCOMES:
Adjusted Therapy Scale (ATI) | Week 1 to Week 11
Addiction Severity Index (ASI) | Week 1 to Week 11
  History and the severity of addiction
Cues of each participant (QSA) | Week 1 to Week 11
Mini International Neuropsychiatric Interview (MINI) | Week 1 to Week 11
  Psychiatric comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Mélina Fatseas, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Bordeaux University Hospital, Bordeaux
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Centre Hospitalier Esquirol, Limoges
  - Centre Hospitalier Universitaire La Réunion, Saint-Denis